CLINICAL TRIAL: NCT05698511
Title: Multivariate Neural and Physiological Correlates of Psychedelic Sub-states: a Within-subjects, Healthy Volunteer Study With Experience-sampling
Brief Title: Neural and Physiological Correlates of Psychedelic Sub-states
Acronym: i2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robin Carhart-Harris, PhD, MA (Other)
Responsible Party: Sponsor-Investigator, Robin Carhart-Harris, PhD, MA, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-35696; 157762 (Other: FDA IND)
Record Dates: First submitted 2022-12-13; First posted 2023-01-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psychedelic Experiences; Neuroimaging; Healthy Volunteers
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Healthy volunteers will receive up to four doses of psilocybin separated from each other by at least one week. The first dosing session will involve 10 mg psilocybin, the remaining three dosing sessions will receive up to 25mg psilocybin.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Multiple dosing of healthy volunteers with up to 25 mg psilocybin separated from each other by at least one week. Participants will be scanned before and after receiving psilocybin on each dosing day. Surveys will be performed on dosing days and after dosing.

SUMMARY:
The main purpose of this study is to gain a better understanding of the distinct mental states and physical reactions that can arise during a psychedelic experience. By repeatedly assessing the same participants in an MRI while under the effects of psilocybin, the investigators want to identify reliable brain and body reactions arising during these psychedelic experiences. It is hoped that this will provide an insight to inspire future research on psilocybin and related psychedelics as well as inform on their therapeutic action. This study will involve up to 12 healthy volunteers with previous psychedelic experience. Participants in this study will be given four doses of psilocybin, with breaks of at least seven days in between dosing visits. The first dosing visit will feature a 10 mg dose of psilocybin, which can be considerate a low to moderate dose, whereas the remaining three dosing visits will feature 25 mg psilocybin, a high dose that is consistent with the dosage chosen for several modern clinical trials with psilocybin. From the initial in-person screening visit to the final follow-up, participants will be in this study for approximately 6-12 weeks and visit the research site 5 times. The first visit will be an in-person screening visit, during which the investigators will assess participants' eligibility to be enrolled. There will be 4 subsequent visits to the scan center for dosing and magnetic resonance imaging (MRI) scanning, and there will be a final remote follow up. Each of the four dosing visits will include four periods of lying within the MRI scanner for scanning, each of these 'in-scanner' sessions will last for ~ 45 minutes. Actual scans, which are also called 'runs' last for ~ 12 mins. During these 'runs', the investigators will ask participants two brief questions about how positive or negative their current experience is every 100 seconds. They will be able to record their answers using a button box which they will be operating with their hand. One day after each dosing visit, the investigators will schedule a phone call with the participant to check how they are doing and perform an informal interview focused on their experience while under the effects of psilocybin.

ELIGIBILITY:
Inclusion Criteria:

* Have had previous experiences with psychedelic substances
* Mentally and physically healthy
* Have had prior experiences with MRI machines (optional but preferred)
* Flexible schedule- able to commit to scans once or twice per week for 4 weeks in a row
* Are between 21 and 70 years of age
* Are fluent in speaking and reading English
* Can swallow pills/capsules
* If able to become pregnant, must be non-lactating, have a negative pregnancy test at study entry and prior to each Experimental Session and must agree to an adequate form of birth control and contraception over the course of the study. Adequate forms of birth control or contraception include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e. condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Not of childbearing potential is defined as documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and/or tubal ligation), permanently sterile by medical device such as Essure, postmenopausal, or male by birth. Contraception applies to males as well as females and male participants must not be planning sperm donation within the study period.
* Able and willing to provide informed consent
* Able and willing to use computers and tablets or phones to enter electronic data
* Agree to inform the investigators within 48 hours of any new or changed medical conditions.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Brain-averaged normalized global signal complexity | Peak effects (120 min post dosing) vs pre-dose
  Signal complexity of brain activity derived from resting-state fMRI

SECONDARY OUTCOMES:
EEG-derived signal complexity of brain activity | Peak effects (120 min post-dose) vs pre-dose fMRI runs
  Measure of brain complexity derived from EEG
Psychological insight | Peak effects (120-min post-dose) vs predose
  Measure of psychological insight

CONTACTS AND LOCATIONS:
Overall Officials: Robin Carhart-Harris, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No